CLINICAL TRIAL: NCT05315700
Title: An Open-Label, Phase 1/2 Study of ORIC-114 as a Single Agent or in Combination With Chemotherapy, in Patients With Advanced Solid Tumors Harboring an EGFR or HER2 Alteration
Brief Title: Study of ORIC-114 in Patients With Advanced Solid Tumors Harboring an EGFR or HER2 Alteration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORIC-114-01
Record Dates: First submitted 2022-03-24; First posted 2022-04-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors
Keywords: EGFR exon 20 insertion mutation; Atypical EGFR mutation; HER2 exon 20 insertion mutation; HER2 amplification/overexpression; NSCLC; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Interval 3+3 dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation and Dose Optimization (Experimental): ORIC-114 dosed orally on a continuous once daily dosing regimen in 28-day cycles.
  Interventions: Drug: ORIC-114
- Combination Dose Escalation (Experimental): ORIC-114 dosed orally on a continuous once daily dosing regimen in 21-day cycles.
  Interventions: Drug: ORIC-114; Drug: Chemotherapy drug

INTERVENTIONS:
Drug: ORIC-114 — ORIC-114 oral daily
Drug: Chemotherapy drug — 21 days for up to 4 cycles
  Other Names: carboplatin and pemetrexed
  Arms: Combination Dose Escalation

SUMMARY:
The purpose of this study is to establish the recommended Phase 2 dose (RP2D) and/or maximum tolerated dose (MTD), safety, pharmacokinetics (PK), pharmacodynamics (PD), and antitumor activity of ORIC-114 as a Single Agent or in Combination with Chemotherapy when administered to patients with advanced solid tumors harboring an EGFR or HER2 alteration.

DETAILED DESCRIPTION:
ORIC-114 is a brain penetrant, selective, orally bioavailable, irreversible small molecule inhibitor designed to target EGFR and HER2 alterations, making it a promising therapeutic candidate for development in patients whose tumors harbor these alterations, including those with CNS metastases.

This is a first-in-human, open-label, single arm, multicenter, dose escalation study of ORIC-114 as a single agent (Part I), followed by dose optimization (Part II) to establish the recommended phase 2 dose (RP2D) and antitumor activity of ORIC-114 in patients with advanced solid tumors harboring an EGFR or HER2 alteration who have exhausted available treatment options. After the optimal RP2D has been determined, Phase 2 will be initiated via protocol amendment to add one or more expansion cohorts of patients with specific tumor types, treatment history, and/or expression of a specific biomarker to evaluate the antitumor activity of ORIC-114.

After completion of Part I dose escalation, Part III, a dose escalation study of ORIC-114 in combination with chemotherapy (carboplatin-pemetrexed) may be initiated to establish the RP2D and/or MTD and antitumor activity for the combination (US sites only).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumor with a documented EGFR or HER2 exon 20 insertion mutation or atypical EGFR mutation as determined by any nucleic acid-based diagnostic testing method, or HER2 amplification/overexpression as determined by an immunohistochemistry (IHC) or an in situ hybridization (ISH) test

  1. Part I Dose Escalation (CLOSED) Any solid tumor with

     * EGFR exon 20 insertion mutation
     * HER2 exon 20 insertion mutation
     * Atypical EGFR mutations (NSCLC only) (Appendix 8)
     * HER2 amplification or overexpression (HER2+)
     * Previously received and progressed on or after available standard therapies and for whom additional standard therapy is considered unsuitable or intolerable
  2. Part I Extension (ONGOING)

     * Cohort IA: Patients with HER2+ breast cancer previously received and progressed on or after available standard therapies and for whom additional standard therapy is considered unsuitable or intolerable
     * Cohort IB: NSCLC patients with EGFR exon 20 insertion mutation previously treated with chemotherapy and amivantamab
     * Cohort IC: Treatment-naïve NSCLC patients with EGFR exon 20 insertion mutation
     * Cohort ID: Treatment-naïve NSCLC patients with EGFR atypical mutations
  3. Part II Dose Optimization (ONGOING): NSCLC patients with

     * Cohort IIA: EGFR exon 20 insertion mutation, patients must have received platinum-based chemotherapy or other chemotherapy regimen if platinum- based chemotherapy was contraindicated. Additionally, patients must be naïve to an EGFR exon 20 targeted agent, ie, must have declined or be ineligible for all available exon 20 targeted therapies with proven benefit
     * Cohort IIB: HER2 exon 20 insertion mutation, patients must have received platinum-based chemotherapy or other chemotherapy regimen if platinum- based chemotherapy was contraindicated. Additionally, patients must be naïve to a HER2 exon 20 targeted TKI
     * Cohort IIC: Atypical EGFR mutation, patients may have received a prior EGFR TKI
* Agreement and ability to undergo pretreatment biopsy
* Measurable disease according to RECIST 1.1
* CNS involvement, which is either previously treated and controlled, or untreated and asymptomatic
* ECOG performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Known EGFR T790M mutation
* Leptomeningeal disease and spinal cord compression

  -- Except if LMD has been reported radiographically on baseline MRI, but is not suspected clinically by the Investigator; the subject must be free of neurological symptoms of LMD
* History of class III or IV congestive heart failure or severe non-ischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months
* Past medical history of interstitial lung disease (ILD), drug induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD
* Known, symptomatic human immunodeficiency virus (HIV) infection
* Known active infection requiring treatment or history of hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients positive for HBsAg but normal HBV DNA level are allowed.
* Active gastrointestinal disease (eg, Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes
* Any other concurrent serious uncontrolled medical, psychological, or addictive conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 12 months
  RP2D as determined by interval 3+3 dose escalation design
Maximum plasma concentration (Cmax) | 28 Days
  PK of ORIC-114
Time of maximum observed concentration (Tmax) | 28 Days
  PK of ORIC-114
Area under the curve (AUC) | 28 Days
  PK of ORIC-114
Apparent plasma terminal elimination half-life (t1/2) | 28 Days
  PK of ORIC-114

SECONDARY OUTCOMES:
Objective response rate (ORR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response (DOR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Clinical benefit rate (CBR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression-free survival (PFS) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Intracranial response rate (CR and/or PR) | 36 months
  Modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Intracranial progression-free survival (PFS) | 36 months
  Modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, MS, Study Director — ORIC Pharmaceuticals
Locations (42):
- United States (17):
  - City of Hope, Duarte, California
  - City of Hope, Huntington Beach, California
  - City of Hope, Irvine, California
  - City of Hope, Long Beach, California
  - University of California, San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health Perlmutter Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Next Oncology, Fairfax, Virginia
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown
  - Peter MacCallum Cancer Centre, Melbourne
  - One Clinical Research, Hollywood Medical Centre, Nedlands
  - Sydney Adventist Health, Sydney
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- The Chinese University of Hong Kong, Shatin, Hong Kong
- Malaysia (5):
  - Sultan Ahmad Shah Medical Centre at International Islamic University Malaysia (IIUM), Kuantan, Pahang
  - Pulau Pinang Hospital, George Town, Pulau Pinang
  - Sarawak General Hospital (SGH), Kuching, Sarawak
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Center (UMMC), Kuala Lumpur
- Medical University of Gdańsk, Gdansk, Poland
- South Korea (8):
  - Chungbuk University Hospital, Cheongju-si
  - National Cancer Center, Goyang-si
  - Catholic University of Korea, St, Vincent Hospital, Gyeonggi-do
  - Gachon University Hospital, Incheon
  - Seoul National Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (3):
  - NEXT Oncology - Barcelona, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - NEXT Oncology - Madrid, Madrid
- National Taiwan University Hospital, Taipei, Taiwan
- The Christie NHS Foundation Trust, Manchester, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No